CLINICAL TRIAL: NCT06130696
Title: Effects of Clamshell Exercises on Pain, Range of Motion and Functions in Athletes With Patellofemoral Pain Syndrome.
Brief Title: Clamshell Exercise in Patellofemoral Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 42663 Anosh Malik
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Clamshell exercises.; Pain; Patellofemoral pain syndrome; Function; Athelete
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clamshell exercise (Experimental): Clamshell exercise
  Interventions: Other: Clamshell exercises
- strengthening exercises with clamshell exercise (Active Comparator): Isometric and muscle strengthening exercises with clamshell exercise.
  Interventions: Other: Isometric and muscle strengthen exercise

INTERVENTIONS:
Other: Clamshell exercises — Group A will receive treatment with Clamshell exercises Change sides and do 3 sets. Total of 6 session were given.
  Arms: Clamshell exercise
Other: Isometric and muscle strengthen exercise — group B will receive simple exercises also with clamshell 10 to 20 times. Change sides and do 3 sets.
  Total 6 session were given
  Arms: strengthening exercises with clamshell exercise

SUMMARY:
Patellofemoral pain syndrome (PFPS), also known as runner's knee, is a common knee condition characterized by pain and discomfort in the front of the knee, specifically around the patella (kneecap) and the surrounding area.

The causes for anterior knee pain are multifactorial like overuse, muscle imbalances abnormal tracking of the patella, biomechanical issues, and improper alignment of the lower limbs. Activities that involve repetitive knee motion, such as running, jumping, squatting, or climbing stairs, can exacerbate the condition . The PFPS may cause aching pain around the front of the knee , especially when sitting for long periods, squatting, or climbing stairs, Pain worsens with activities that involve bending the knee, popping or grinding sensation in the knee and swelling or inflammation around the knee in some cases.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) leads to pain and restricted activities in athletes. There are many remedies used to tackle this problem like Physical therapy, Orthotics or shoe inserts, Patellar taping or bracing, RICE therapy, Nonsteroidal anti-inflammatory drugs (NSAIDs) and in some cases, corticosteroid injections are administered to reduce pain and inflammation. A randomized control trial will be conducted at Pakistan Sports Board Lahore through nonprobability convenience sampling technique on 38 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A and group B. Group A will receive treatment with Clamshell exercises and group B will receive simple exercises for a period of six weeks. Side-lying clam exercises include lying down on one side on an exercise mat placing the head on arm and top leg/foot on lower leg/foot. Then lift the top leg towards ceiling and lower it again upto 10 to 20 times. Change sides and do 3 sets. Outcome measures such as range of motion will be measured by goniometer and pain by NPRS Scale, Visual analogue Scale and Kujala Patellofemoral pain score and the functional status will be measured with functional mobility test and physical performance testing. Patellar grind test for knee pain will also be performed at start and end to see the effectiveness of Clamshell exercise in athletes.

Data will be analyzed using SPSS software version 21. After assessing normality of data, it will be decided either parametric or non-parametric test will be used within a group or between two groups. Effectiveness of clamshell exercises will be analyzed by comparison in individuals with PFPS.The significance of this study lies in evaluating the effectiveness of clamshell exercises of hip muscles on PFP. The clamshell exercise can be beneficial for individuals with PFPS as part of a comprehensive rehabilitation program as it primarily targets the hip abductor muscles and indirectly contributes to improving knee stability and addressing muscle imbalances that can affect PFPS.

Based on the above stated literature review focusing on PFPS, its effects and remedies, we can conclude that athletes with PFPS shows signs of improvement when re-engaged in training activities. Also Clamshell exercises have wide impact to address muscles and knee problems, so there is a dire need to fill a research gap and study the impact of these exercises on PFPS with special focus on athletes facing the pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients have at least three months history of peri- or retropatellar pain with worst pain intensity during previous week of VAS 3 or more.
* Players with complain of knee pain.
* Individual having pain during compression of the patella, palpation of the patellar facets

Exclusion Criteria:

* Any degenerative changes of the knee or hip.
* History of patellar dislocation.
* Evidence of edema, Osgood-Schlatter disease or Sinding-Larsen-Johanssen syndrome, patellar -tendinopathy, chondral injury, osteoarthritis.

Joint or muscle injuries in the hip, lumbar pain, sacroiliac pain.

-Patients who previously received surgical treatment in the knee or hip joints, and bilateral complaint of anterior knee pain

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Kujala patellar scale. (Pain ) | 4th day
  diagnostic tool that aims to assess the severity of symptoms and physical limitations in patients with patellofemoral pain syndrome (PFPS). 13-item self-questionnaire that assesses to limitation physical activities and symptoms that are known to correlate with anterior knee pain syndrome.
  This scle consist 0 - 100 score. Less than 90 shows physcial limitation or pain at patellar site. While 98 or 100 shows good knee with no pain or limitation.
Goniometer. (ROM) | 4th day
  Goniometer is used to measure the range of motion of joint. For knee joint, flexion ranges between 0-135º and extension ranges between 135-0º.
Functional mobility test ( physical activity / function) | 4th day
  Functional mobility test: Functional movement screen (FMS) is an evaluation tool for whom movement is a key part of exercise. FMS consists of 7 movement pattern and 3 three clearing tests assess pain for shoulder rotation motions, trunk extension, and trunk flexion. The FMS is scored on an ordinal scale, with 4 possible scores ranging from 0 to 3. 'Zero' refers if the individual has pain during any part of the movement. '1' represents that the person is unable to complete the movement pattern, '2' represents the ability to complete the movement with compensation and '3' refers that the person completes the movement without compensation

SECONDARY OUTCOMES:
Manual muscle testing. | 4th week
  Manual muscle testing is an assessment of muscle strength .The score of '0' represents no activity. '1' represents trace contractile activity but no resulting movement. '2' represents full ROM only in horizontal plane. '3' represents full ROM against the effect of gravity. '4' represents full ROM against gravity and test position is held under minimum resistance. '5' represents full ROM against gravity and test position is held under maximum resistance.
  Grade 5 shows good muscle power.
Numeric pain rating scale. | 4th week
  Numeric pain rating scale is 11-point scale ranges from "0" no pain to "10' worst imaginable pain.
Visual analogue scale | 4th week.
  Visual analogue scale measures pain that ranges across a continuum from none to an extreme amount of pain. VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient mark

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boling M, Padua D, Marshall S, Guskiewicz K, Pyne S, Beutler A. Gender differences in the incidence and prevalence of patellofemoral pain syndrome. Scand J Med Sci Sports. 2010 Oct;20(5):725-30. doi: 10.1111/j.1600-0838.2009.00996.x. PMID 19765240
- [Background] Robinson RL, Nee RJ. Analysis of hip strength in females seeking physical therapy treatment for unilateral patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2007 May;37(5):232-8. doi: 10.2519/jospt.2007.2439. PMID 17549951
- [Background] Pereira PM, Baptista JS, Conceicao F, Duarte J, Ferraz J, Costa JT. Patellofemoral Pain Syndrome Risk Associated with Squats: A Systematic Review. Int J Environ Res Public Health. 2022 Jul 28;19(15):9241. doi: 10.3390/ijerph19159241. PMID 35954598
- [Background] Fang B, Kim YH, Choi MY. Effects of High-Intensity Aquatic or Bicycling Training in Athletes with Unilateral Patellofemoral Pain Syndrome. Int J Environ Res Public Health. 2022 Apr 13;19(8):4675. doi: 10.3390/ijerph19084675. PMID 35457543
- [Background] Al-Hakim W, Jaiswal PK, Khan W, Johnstone D. The non-operative treatment of anterior knee pain. Open Orthop J. 2012;6:320-6. doi: 10.2174/1874325001206010320. Epub 2012 Jul 27. PMID 22896779
- [Background] Campbell SA, Valier AR. The Effect of Kinesio Taping on Anterior Knee Pain Consistent With Patellofemoral Pain Syndrome: A Critically Appraised Topic. J Sport Rehabil. 2016 Aug;25(3):288-93. doi: 10.1123/jsr.2014-0278. Epub 2015 May 6. PMID 25946512